CLINICAL TRIAL: NCT07081659
Title: On-demand Silodosin 4mg vs Dapoxetine 60mg in the Treatment of Primary Premature Ejaculation
Brief Title: On-demand Silodosin 4mg vs Dapoxetine 60mg in Treatment of Primary Premature Ejaculation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Hussein Shaher, assisstant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ms13-3-2024
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Premature (Early) Ejaculation
Keywords: premature ejaculation; sexual function; ejaculatory profile; latency time
MeSH Terms: conditions — Premature Birth; Premature Ejaculation | interventions — dapoxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): sildosin 4mg
  Interventions: Drug: sildosin 4mg
- group B (Active Comparator): dapoxetine 60mg
  Interventions: Drug: dapoxetine 60mg

INTERVENTIONS:
Drug: sildosin 4mg — ondemand sildosin 4mg
  Arms: group A
Drug: dapoxetine 60mg — ondemand dapoxetine 60mg
  Arms: group B

SUMMARY:
Both Silodosin 4 mg and Dapoxetine 60 mg significantly improved IELT and sexual function scores in primary PE patients. However, Silodosin exhibited a more favorable tolerability profile with fewer side effects, making it a safer, clinically effective alternative.

DETAILED DESCRIPTION:
Dapoxetine 60 mg, the initial FDA-approved on-demand treatment for PE, which is a selective serotonin reuptake inhibitor (SSRI) . However, Silodosin 4 mg, an α1-adrenoceptor antagonist, has emerged as a promising alternative, particularly for patients dissatisfied with Dapoxetine . This investigation is designed to evaluate the efficacy and tolerability of Silodosin 4mg and Dapoxetine 60mg in the treatment of primary premature ejaculation.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual male
* Sexually active
* Aged 25 to 65 years old.
* Primary premature ejaculation (IELT < 1 minute)
* They had experienced PE for a minimum of 6 months

Exclusion Criteria:

* Patients with a history of diabetes or
* Uncontrolled hypertension (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg) was precluded from the study.
* Anatomic abnormalities of the penis or genital region,
* Erectile dysfunction,
* Chronic prostatitis,
* Psychological disorder
* Patients on anti-psychotic drugs.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patients in heterosexual relation
Enrollment: 95 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Intravaginal ejaculatory Latency time | 2 months
  changes in latency time

SECONDARY OUTCOMES:
side effects | 2 months
  any side effects were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Benha faculty of medicine, urology department, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
it will be shared upon request
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT07081659/Prot_SAP_000.pdf